CLINICAL TRIAL: NCT07215091
Title: Effectiveness and Implementation of a Brief Motivational Intervention to Increase Physical Activity for World Trade Center Health Program Cancer Survivors
Brief Title: Testing a Brief Motivational Intervention to Increase Physical Activity for Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Pamela Ginex, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB2024-00344; 5R21OH012630-02 (NIH)
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: World Trade Center Health Program
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Motivational Intervention:
  The intervention group will receive a 3-component motivational intervention based on the Theory of Planned Behavior in addition to an enhanced standard of care. The components of the intervention include motivational interviewing (MI); mobile health monitoring; and action planning.
  At the initial visit, following baseline data collection, the clinician will use MI to build a positive attitude towards physical activity (PA). Next, they will discuss why and how to use Fitbit to monitor steps per day. The last component of the intervention includes action planning to design a PA program that fits their abilities and lifestyle. Following the in-person baseline visit, participants will be called approximately every 2 weeks during the 3-month intervention period. During these calls, the action plan will be reviewed and updated, and their step count reviewed.
  Interventions: Behavioral: Brief Motivational Intervention
- Wait List Control (Active Comparator): Wait List Control:
  The control group will receive a Fitbit and advice to continue their normal physical activity. At the end of 3 months, the wait-list control group will be seen in the clinic for the motivational intervention which will be the same as the intervention group. They will return to the clinic at the end of the study (6 months) for final data collection. Participants in the wait list control group will use the Fitbit for the full 6 months of the study, during the 3 month waiting period and the 3 month intervention.
  Interventions: Behavioral: Brief Motivational Intervention

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — The study includes a 3-component motivational intervention based on the Theory of Planned Behavior. The components include motivational interviewing (MI); mobile health monitoring; and action planning.
  MI is used to build a positive attitude towards physical activity (PA). Mobile health monitoring will be conducted with a Fitbit to monitor steps per day. The last component of the intervention includes action planning to design a PA program that fits their abilities and lifestyle. The research team will develop a PA grid that includes aerobic, strength, and flexibility PA options. The PA grid provides an opportunity to personalize the action plan by choosing from a 'menu' to match interests. Following the in-person baseline visit, participants will be called approximately every 2 weeks (4-5 phone contacts) during the 3-month intervention period to review and update their action plan.

SUMMARY:
The goal of this study is to test a brief motivational intervention to increase physical activity in a group of cancer survivors who are participants in the World Trade Center Health Program.

DETAILED DESCRIPTION:
The World Trade Center Health Program (WTCHP) tracks the ongoing health and well-being of over 91,000 first responders and people who lived and worked near the World Trade Center. Research has established that WTCHP members are at higher risk for a constellation of health conditions, including cancer. Cancer survivors, the focus of this study, are at risk for physical and functional impairment. As WTCHP members with cancer age, developing pragmatic interventions to mitigate physical decline is an important next step in a coordinated program of care and research in this vulnerable population. Physical activity (PA) interventions are strong candidates for investigation, given that physical inactivity in WTCHP members has been correlated with respiratory illness, poor sleep, and PTSD. PA has many health benefits, yet interventions to support PA are not routinely incorporated into clinical practice. Evidence-based guidelines recommend PA counseling in clinical care and health professionals believe they should be doing this. However, a gap remains in implementing PA interventions at the point of care. This study will test an evidence-based motivational intervention to initiate and maintain PA among WTCHP particpatants with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the World Trade Center Health Program
* History of cancer, completed treatment
* Ability to be physically active (at minimum be able to walk slowly)

Exclusion Criteria:

* Participants receiving active cancer treatment (excluding hormonal therapy);
* Late-stage cancer (metastatic);
* Inability to follow the scheduled visits;
* Women who are pregnant
* Patients who would not be safe exercising without medical supervision (ECOG score of 3, significant comorbidities, unable to even walk slowly)
* Inability to speak and read English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-01-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity | Baseline to end of study (6 months)
  The primary outcomes will be measured with Fitbit data. Fitbit software allows classification of each minute as being in sedentary, light, moderate, or vigorous activity, and provides metabolic equivalents (METs) for each minute. Positive changes in levels of physical activity will be determined by a 25% increase in MVPA from baseline to end of intervention. This estimation is based on a systematic review of motivational physical activity interventions in cancer survivors (Takemura, 2024). This change in outcome measure is well justified and sensitive to small changes in activity.

SECONDARY OUTCOMES:
Quality of Life (SF-20) | Baseline to end of study (6 months)
  SF-20 includes 20 quality-of-life statements that are well validated and reliable. The survey measures health across 6 domains: physical functioning (6 questions), role functioning (2 questions), social functioning (1 question), mental health (5 questions), health perceptions (5 questions), and pain (1 question). The total score will be used to measure quality of life and the physical functioning domain score will be used to subjectively measure physical functioning. Higher scores indicate better health.
Sleep (PROMIS Sleep SF) | Baseline to end of study (6 months)
  Sleep will be measured with the PROMIS Sleep Disturbance short form, a 6-item scale that assesses sleep quality and satisfaction with sleep on a five-point Likert scale. The scale is reliable and valid and correlates strongly with longer forms. Higher scores indicate more sleep disturbance.
Fatigue (PROMIS Fatigue SF) | Baseline to end of study (6 months)
  Fatigue will be measured with the PROMIS Fatigue short form. This scale includes 8 items related to fatigue and the impact of fatigue on day-to-day life. The form has good reliability (0.88) and validity (.60 -.85) across different groups and has been used across diverse clinical populations. Higher scores indicate more fatigue.
Physical Functioning (Short Physical Performance Battery) | Baseline to end of study (6 months)
  Physical function will be derived from performance on the Short Physical Performance Battery (SPPB). The SPPB consists of 3 components: balance (side-by-side, semi-tandem, and tandem positions held for 10 seconds unassisted), gait speed (amount of time to walk a four-meter course at a typical pace), and repetitive chair stand (amount of time to rise from a chair unassisted 5 consecutive times). Each component is rated on a 4-point scale based on the ability and amount of time necessary to complete each task. SPPB ≥10 indicated scores in the normal range, whereas a score of ≤9 indicated functional impairment (further stratified into mild (7-9) vs moderate (4-6) to severe (≤3)). Grip strength will be measured by using a standard dynamometer and assessed from a single 3-s maximal grip effort of the right- and left-side arms. Decreased grip strength has been strongly associated with a range of adverse health outcomes.
Post traumatic stress disorder (PCL-5) | Baseline to end of study (6 months)
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report questionnaire that assesses Post-Traumatic Stress Disorder (PTSD) symptoms on a 5-point Likert scale, with total scores ranging from 0 to 80. Symptoms are grouped into four clusters corresponding to DSM-5 PTSD criteria, and scoring involves summing item responses to calculate a total score or to identify minimum symptom endorsement for a provisional diagnosis. Higher scores indicate more severe PTSD symptoms, with scores of 31-33 or above generally considered clinically significant and potentially indicative of PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided